CLINICAL TRIAL: NCT00388011
Title: Randomized, Double-Blind, Placebo and Comparator-Controlled, Dose-Response Trial of the Efficacy and Safety of Intranasal Morphine, Intravenous Morphine and Placebo in Patients With Moderate to Severe Pain Following Orthopedic Surgery
Brief Title: Efficacy and Safety of Intranasal Morphine for Pain After Bunion Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Javelin Pharmaceuticals (Industry)
Responsible Party: Amy Cohen/Director, Clinical Operations, Javelin Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MOR-002
Record Dates: First submitted 2006-10-12; First posted 2006-10-13 (Estimated); Last update posted 2008-01-14 (Estimated); Status verified 2008-01

CONDITIONS: Hallux Valgus
Keywords: Post surgical pain; Bunionectomy; Hammer Toe Syndrome; Morphine
MeSH Terms: conditions — Hallux Valgus; Pain, Postoperative; Hammer Toe Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (Experimental): Intranasal morphine 3.75 mg
  Interventions: Drug: Intranasal Morphine (MNS075) 3.75 mg
- 2 (Experimental): Intranasal morphine 7.5 mg
  Interventions: Drug: Intranasal morphine (MNS075) 7.5 mg
- 3 (Experimental): Intranasal morphine 15 mg
  Interventions: Drug: Intranasal morphine (MNS075) 15 mg
- 4 (Experimental): Intranasal morphine 30 mg
  Interventions: Drug: Intranasal morphine (MNS075) 30 mg
- 5 (Active Comparator): Intravenous morphine 7.5 mg
  Interventions: Drug: Intravenous Morphine 7.5 mg
- 6 (Placebo Comparator): Intranasal placebo
  Interventions: Drug: Intranasal placebo

INTERVENTIONS:
Drug: Intranasal Morphine (MNS075) 3.75 mg — Intranasal Morphine (MNS075) 3.75 mg
  Arms: 1
Drug: Intravenous Morphine 7.5 mg — Intravenous Morphine 7.5 mg
  Arms: 5
Drug: Intranasal morphine (MNS075) 7.5 mg — Intranasal morphine (MNS075) 7.5 mg
  Arms: 2
Drug: Intranasal morphine (MNS075) 15 mg — Intranasal morphine (MNS075) 15 mg
  Arms: 3
Drug: Intranasal morphine (MNS075) 30 mg — Intranasal morphine (MNS075) 30 mg
  Arms: 4
Drug: Intranasal placebo — Intranasal placebo
  Arms: 6

SUMMARY:
Study designed to evaluate the efficacy and safety of Intranasal (IN) Morphine Nasal Spray (MNS075) 3.75 mg, 7.5 mg, 15 mg, and 30 mg, intravenous (IV) morphine 7.5 mg, or IN placebo in patients with moderate to severe post-surgical pain following orthopedic surgery. After initial dosing, up to six (6) doses of IN MNS075 7.5 mg or 15 mg for up to twenty-four (24) hours will be evaluated. The rescue dose remained the same for each.

DETAILED DESCRIPTION:
Diagnosis and Main Criteria for Inclusion:

Healthy adult patients (18 to 76 years old), who scored PS-1 to PS-3 according to the American Society of Anesthesiologists Physical Status Classification System, requiring primary, unilateral, first metatarsal bunionectomy surgery alone or with ipsilateral hammertoe repair without additional collateral procedures.

ELIGIBILITY:
Inclusion Criteria:

* Requires primary unilateral first metatarsal bunionectomy surgery alone or with ipsilateral hammertoe repair under regional anesthesia. The patient requires collateral orthopedic surgical procedures other than ipsilateral hammertoe repair may not be enrolled into the study.
* 18 years of age or older
* Moderate to severe pain within eight (8) hours following completion of the required bunionectomy surgery

Exclusion Criteria:

* Allergy to shellfish
* Signs of nasal congestion, nasal polyps, mucosal lesions of the nostrils, postnasal drip of any etiology or any clinically significant nasal pathology that may affect the absorption of study medication or the assessment of safety.
* Chronic respiratory insufficiency such that treatment with an opioid analgesic is contraindicated

Additional Inclusion/Exclusion Criteria May Apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2005-01; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
VAS Total Pain Relief 0-4 hours (TOTPAR4) | 4 hours

SECONDARY OUTCOMES:
Other measures of pain relief | Several time points

CONTACTS AND LOCATIONS:
Overall Officials: Douglas G Stoker, DPM, Principal Investigator — Jean Brown Research